CLINICAL TRIAL: NCT07014501
Title: Study on the Correlation Mechanism and Application of Genetic Susceptibility, Hemoglobin Adaptation Changes, and Extubation Success Rate in Stroke Patients With Tracheotomy at Different Altitudes
Status: Recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Department of rehabilitation medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Other Study IDs: Shen-PJ-Ke-2025-94
Record Dates: First submitted 2025-05-19; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Stroke; Tracheotomy Patients
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High altitude group: High altitude stroke patients with tracheotomy.
  Interventions: Other: High altitude
- Medium altitude group: Stroke patients with moderate altitude combined with tracheotomy.
  Interventions: Other: Low altitude group
- Low altitude group: Low altitude stroke patients with tracheotomy.
  Interventions: Other: Medium altitude

INTERVENTIONS:
Other: High altitude — Altitude above 3500 meters.
  Groups: High altitude group
Other: Medium altitude — Altitude between 3500 meters and 1500 meters.
  Groups: Low altitude group
Other: Low altitude group — Altitude below 1500 meters.
  Groups: Medium altitude group

SUMMARY:
Patients with brain injuries caused by various reasons often need tracheotomy to improve breathing, but this procedure can cause the air to lose its nasal regulation, increase the risk of lung infections, and reduce their quality of life. Tracheal extubation is crucial for patient recovery. Environmental factors in high-altitude areas have a significant impact on human cardiovascular function, including changes in blood oxygen caused by low oxygen environments and cardiovascular adaptability of long-term residents. There is limited research on the impact of high altitude on the success rate of tracheal extubation in brain injury. The research team conducted a retrospective study on 501 patients who underwent tracheotomy at the Second Affiliated Hospital of Kunming Medical University and found that high GCS scores and hemoglobin concentrations were beneficial for extubation. The increase in hemoglobin concentration among high-altitude residents may be an adaptive response to hypoxia, and the research team speculates that this may become a protective factor for successful extubation. However, some argue that altitude sickness and adaptive genetic changes may counteract each other. Simonson's team found that the decline of hemoglobin concentration in Tibetans was related to specific gene expression, indicating that the genetic adaptability of high altitude residents had a unique relationship with hemoglobin concentration. Therefore, the research team speculates that people living in highlands for a long time are more adaptable to hypoxic environments than those living in lowlands. Under severe stress (hypoxia), people living in highlands for a long time may have lower sensitivity to pulmonary blood flow redistribution or oxygen delivery compared to those living in lowlands. This study is a multicenter observational study, with sub centers listed as follows: Jiangchuan District People's Hospital, Huaning County People's Hospital, Baoshan Second People's Hospital, Huize County People's Hospital, Mengla County People's Hospital, Tonghai County People's Hospital, Jinghong City First People's Hospital, Xuanwei City First People's Hospital, Qiubei County People's Hospital, Fengqing County People's Hospital, Weixin County People's Hospital, Yulong County People's Hospital, Yanshan County People's Hospital, Xundian County People's Hospital, Shizong County People's Hospital, Luxi County People's Hospital, Yunnan Province Northeast Yunnan Central Hospital, Luoping County People's Hospital, Xinping County General Hospital, Suijiang County People's Hospital, Nanhua County Hospital, Guangnan County People's Hospital County People's Hospital, Jianshui County People's Hospital, Simao District People's Hospital of Pu'er City, Funing County People's Hospital, Xinping County Traditional Chinese Medicine Hospital Xundian County First People's Hospital and Jingdong County People's Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Hospitalized patients in the rehabilitation department with acute non-traumatic ischemic stroke, intracerebral hemorrhage, or subarachnoid hemorrhage requiring tracheostomy.
3. Hemodynamic stability: Systolic blood pressure maintained between 90-160 mmHg, diastolic blood pressure between 60-100 mmHg, respiratory rate between 12-30 breaths/min, heart rate between 60-120 beats/min, body temperature between 36.5°C-38.5°C, and arterial oxygen saturation (SaO₂) consistently >90% at admission and prior to tracheostomy.
4. Glasgow Coma Scale (GCS) score of 5-15 at assessment.
5. Tracheostomy performed within 24-72 hours after stroke onset.
6. Peripheral blood hemoglobin concentration at admission within specified ranges (male: 120-180 g/L; female: 110-160 g/L).
7. Signed informed consent provided by the patient or legal guardian.

Exclusion Criteria:

1. History of severe cardiopulmonary dysfunction (e.g., chronic obstructive pulmonary disease, cor pulmonale, coronary artery disease, cardiomyopathy) with New York Heart Association (NYHA) functional class III or IV, or recent (within 6 months) acute myocardial infarction or unstable angina.
2. Diagnosis of advanced malignancy (life expectancy <6 months) with ongoing chemotherapy, radiotherapy, or palliative care.
3. Severe hepatic or renal insufficiency (e.g., decompensated cirrhosis, chronic renal failure requiring long-term dialysis).
4. Uncontrolled endocrine disorders (e.g., thyrotoxic crisis, myxedema coma, diabetic ketoacidosis, hyperosmolar hyperglycemic state).
5. Coagulation disorders:

   * Congenital or acquired coagulopathies (e.g., hemophilia, vitamin K deficiency, coagulation factor deficiency due to severe liver disease, antiphospholipid syndrome).
   * Active anticoagulation therapy (e.g., warfarin with INR >3.0, heparin with APTT exceeding twice the upper limit of normal) unadjustable to a safe range within 72 hours.
6. Major surgery within 3 months (e.g., cardiac, abdominal, or orthopedic surgery).
7. Severe chest trauma (e.g., multiple rib fractures, pneumohemothorax) or abdominal trauma (e.g., liver/spleen rupture, intestinal perforation) within 1 month prior to stroke onset, with incomplete recovery.
8. Active uncontrolled infection at admission (e.g., pneumonia, urinary tract infection, intracranial infection, sepsis) defined by:

   * Temperature >38.5°C persisting >24 hours.
   * Elevated white blood cell count, increased neutrophil percentage, and clinical signs of infection.
   * Positive bacterial cultures (blood, sputum, urine).
9. Recent (within 1 week) exposure to infectious diseases (e.g., travel to epidemic areas, contact with confirmed cases) with suspected latent or active infection.
10. History of neurodegenerative diseases (e.g., Parkinson's disease, Alzheimer's disease) or motor neuron disorders (e.g., amyotrophic lateral sclerosis).
11. Congenital neurological developmental abnormalities (e.g., hydrocephalus, cerebral palsy).
12. Severe uncontrolled psychiatric disorders (e.g., schizophrenia, major depressive disorder, bipolar disorder) impairing daily function or treatment adherence.
13. Cognitive impairment (e.g., dementia) with Mini-Mental State Examination (MMSE) score <10.
14. Pregnancy or lactation.
15. Hypersensitivity or contraindications to study-related drugs or procedures (e.g., allergy to tracheostomy tube materials, antibiotic allergies without alternatives).
16. Inability to complete follow-up or required tests (e.g., geographical barriers, unreliable contact information).
17. Non-compliance of the patient or family members with the study protocol.
18. Failure to obtain informed consent.
19. Participation in other interventional clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls hospitalized patients aged 18-75 with acute non-traumatic ischemic stroke, intracerebral hemorrhage, or subarachnoid hemorrhage requiring tracheostomy, stratified by long-term residence altitude: high (>3500m), medium (1500-3500m), and low (<1500m). Target sample: 717 participants (20% attrition). Participants will be recruited from the Rehabilitation Medicine Department of the Second Affiliated Hospital of Kunming Medical University and 27 participating centers. Ethics-approved with written consent and data confidentiality.
Sampling Method: Non-Probability Sample
Enrollment: 717 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-29 (Estimated)

PRIMARY OUTCOMES:
Tracheostomy extubation | Through study completion, an average of 1 year.
  The outcome measure is the success of tracheostomy tube extubation in stroke patients. Successful extubation is defined as extubation of the tracheal tube as planned and not reintubated during subsequent treatment, and survival within 7 days of extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Electroencephalography, Kunming, Yunnan, China